CLINICAL TRIAL: NCT06900894
Title: Effectiveness of Platelet-Rich Fibrin and Elastic Bandaging on Postoperative Pain, Edema, and Recovery Following Impacted Molar Surgery: A Randomized Clinical Trial
Brief Title: Effects of Platelet-Rich Fibrin and Kinesio Taping on Postoperative Recovery in Oral Surgery
Acronym: PRFKTOralSur
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, züleyha başar karakuzu, DDS, Oral and Maxillofacial Surgeon, Mustafa Kemal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRF_KT2025; Ethics Committee No. (Registry Identifier: Hatay Clinical Research Ethics Committee - 2023/03)
Record Dates: First submitted 2025-03-17; First posted 2025-03-28 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Impacted Third Molar Tooth; Postoperative Pain; Postoperative Edema
Keywords: Impacted third molar; elastic bandage; platelet-rich fibrin; postoperative pain; quality of life; Postoperative Edema
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: This study follows a parallel assignment model in which participants are randomly allocated into three groups: Platelet-Rich Fibrin (PRF), Kinesio Taping, and Control. Each group receives a distinct intervention to evaluate the effectiveness of these non-pharmacological approaches in managing postoperative pain, edema, and recovery following impacted third molar surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PRF Group (Experimental): Participants in this group received Platelet-Rich Fibrin (PRF) applied to the extraction socket following impacted third molar surgery. PRF was prepared using a centrifugation protocol and placed into the surgical site.
  Interventions: Biological: Platelet-Rich Fibrin (PRF)
- Kinesio Taping Group (Experimental): Participants in this group received Kinesio Taping applied postoperatively. The elastic therapeutic tape was applied to the masseter and submandibular region following a standardized taping protocol.
  Interventions: Device: Kinesio Taping
- Control Group (Other): Participants in this group received standard postoperative care, including routine pain management and wound care, without additional interventions.
  Interventions: Other: Standard Postoperative Care

INTERVENTIONS:
Biological: Platelet-Rich Fibrin (PRF) — PRF was prepared using a centrifugation protocol and applied to the extraction socket.
  Arms: PRF Group
Device: Kinesio Taping — Kinesio Tape was applied postoperatively to the masseter and submandibular region.
  Arms: Kinesio Taping Group
Other: Standard Postoperative Care — Patients in the control group received standard postoperative care.
  Arms: Control Group

SUMMARY:
This study investigates the effectiveness of Platelet-Rich Fibrin (PRF) and Kinesio Taping in reducing postoperative pain, edema, and improving recovery following impacted third molar surgery. A prospective, randomized clinical trial was conducted with 44 patients aged 18-35 years. Patients were assigned to three groups: (1) PRF applied locally to the extraction socket, (2) Kinesio Taping applied postoperatively and removed on the third day, and (3) a control group receiving standard postoperative care. Postoperative outcomes were assessed on days 3 and 7, including pain levels, edema, and quality of life. This study aims to evaluate PRF and Kinesio Taping as non-pharmacological adjuncts in oral and maxillofacial surgery.

DETAILED DESCRIPTION:
This study investigates the effectiveness of Platelet-Rich Fibrin (PRF) and Kinesio Taping in postoperative management following impacted mandibular third molar surgery. Postoperative complications, such as pain and edema, are commonly observed and may impact patient comfort and recovery. This study aims to evaluate the feasibility of two non-pharmacological approaches-PRF and Kinesio Taping (Elastic Bandaging)-in postoperative care.

A total of 44 patients aged 18-35 years participated in this prospective, randomized clinical trial. Patients were assigned to one of three groups:

PRF Group: Platelet-rich fibrin (PRF) was applied locally into the extraction socket.

Kinesio Taping Group: An elastic bandage was applied postoperatively to the surgical area and removed on the third day.

Control Group: Standard postoperative care was provided with no additional intervention.

Postoperative evaluations were conducted on the 3rd and 7th days. The measured parameters included:

Edema: Measured using anthropometric techniques.

Pain: Assessed with the Numerical Rating Scale (NRS).

Quality of Life: Evaluated using the Oral Health Impact Profile-14 (OHIP-14).

This study aims to assess the feasibility of PRF and Kinesio Taping in postoperative management.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-35 years
* Systemically healthy individuals
* Non-smokers
* No psychological disorders
* Preoperative pain level between 0-3 on the Numerical Rating Scale (NRS)
* No preoperative edema in the surgical area
* Impacted mandibular third molars classified as Class 1 or 2, Level B, and mesioangular according to the Pell-Gregory classification
* Signed an informed consent form

Exclusion Criteria:

* Under 18 or over 35 years old
* Presence of chronic or systemic diseases
* Pregnant or breastfeeding patients
* Surgical duration exceeding 45 minutes
* Smokers
* Patients requiring prophylactic antibiotics due to systemic health conditions
* Patients who did not meet the study criteria or did not sign the informed consent form

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-05-21 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain Assessment (NRS) | Preoperative day 1, postoperative days 3 and 7
  The pain intensity of the patients will be assessed using the Numerical Rating Scale (NRS) on preoperative day 1 and postoperative days 3 and 7.
  On this scale: 0 indicates no pain, 10 indicates the worst imaginable pain. Before the procedure, patients were informed about the scale and instructed to rate their pain intensity accordingly.
Postoperative Facial Swelling Assessment | Preoperative day 1, postoperative days 3 and 7
  Swelling will be evaluated using anthropometric measurement techniques on preoperative (surgery day), postoperative days 1, 3, and 7.
  Measurement methods:
  Lateral canthus-gonion distance (distance from the outer corner of the eye to the mandibular angle) Commissure-tragus distance (distance from the oral commissure to the midpoint of the tragus) All measurements were performed using a flexible ruler, and the results were recorded in millimeters.
Oral Health Impact Profile-14 (OHIP-14) Score | Postoperative days 3 and 7
  The quality of life of the patients will be assessed using the OHIP-14 questionnaire on postoperative days 3 and 7.
  OHIP-14 consists of 14 standardized items, each rated on a scale from 0 to 4. Total scores range from 0 to 56, with higher scores indicating worse quality of life.
  This scale was used to evaluate the impact of postoperative complications on patients' quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: züleyha başar karakuzu, DDS, Principal Investigator — Mustafa Kemal University
Locations (1):
- Hatay Mustafa Kemal University, Faculty of Dentistry, Hatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) collected during the study will not be shared due to confidentiality and ethical considerations. Data will only be used for statistical analysis and publication purposes in an aggregated and anonymized form.